CLINICAL TRIAL: NCT04409678
Title: Influence of Physical Activity on Preterm Birth for Women With Cervical Dynamics
Brief Title: Physical Activity and Preterm Birth With Cervical Dynamics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Yakira, Dr Izaik Yakira, Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0112-19-womc
Record Dates: First submitted 2020-05-26; First posted 2020-06-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- activity (Experimental)
  Interventions: Behavioral: activity
- bed rest (No Intervention)

INTERVENTIONS:
Behavioral: activity — physical activity
  Arms: activity

SUMMARY:
this RCT is designed to investigate the influence of physical activity on the risk f preterm birth for women with cervical dynamics.

ELIGIBILITY:
Inclusion Criteria:

pregnant women between 24-34 weeks of gestation singleton cervical length<25 mm willing to download an application which traces physical activity on medical indication for reducing activity

Exclusion Criteria:

refusal to participate medical advise to minimize activity (symphysiolysis) maternal morbidity fetal compromise vaginal bleeding rapture of membranes severe preeclampsia twins pregnancy

-

Ages: 18 Years to 54 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-05-26 (Actual); Primary Completion 2021-05-26 (Estimated); Study Completion 2021-05-26 (Estimated)

PRIMARY OUTCOMES:
preterm birth | assessed from recruitment to delivery
  birth prior to 37 weeks of gestation

CONTACTS AND LOCATIONS:
Locations (1):
- edith wolfsom MC, Holon, Israel